# A MEDICAL RESEARCH COUNCIL (MRC)/UGANDA VIRUS RESEARCH INSTITUTE (UVRI)/LONDON SCHOOL OF HYGIENE AND TROPICAL MEDICINE (LSHTM) UGANDA RESEARCH UNIT COLLABORATIVE STUDY

# PROTOCOL VERSION 7.0

12 Jan 2019

Study title: Improving uptake and adherence to HIV prevention services with PrEP and HIV self testing for HIV negative high risk young women aged 15-24 in Kampala, Uganda

Short title: The POPPi (Prevention on PrEP) study

Sponsor: NIH / National Institute of Mental Health (NIMH)

Grant # MH114523-01

#### NAMES OF APPLICANTS AND COLLABORATING INSTITUTIONS

Rachel L King, Study PI UCSF 550 16th Street, 3rd Floor San Francisco, CA 94158-1224 USA

Tel: +256 785304516

E-mail: rach@vtx.ch / rachel.king@ucsf.edu

Lisa Butler,—Sub-grantee PI Institute for Collaboration on Health,

Intervention, and Policy University of Connecticut 2006 Hillside Road, Unit 1248 Storrs, CT 06269-1248 Tel: +1 (617) 500-8209

Email: Lisa.Butler@uconn.edu

Andrew Abaasa, Co-Investigator MRC/UVRI/LSHTM Uganda Research Unit Box 49, Entebbe, Uganda Tel: +256712976987 Email: andrew.abaasa@mrcuganda.org

Project Role: Statistician

Jaco Homsy, Co-Investigator
UCSF Site Investigator
MU-JHU, Old Mulago Hill Rd
Kampala, Uganda
Tel: +256 772747097
E-mail: jaco251099@vtx.ch/jaco.homsy@ucsf.edu

NIMH Program Officer: Susannah Allison, PhD 5601 Fishers Lane, Room 9E26 Rockville, MD 20852, USA

Tel: +1-240-627-3861Tel: +1-301-443-3034

E-mail: allisonsu@mail.nih.gov

Janet Seeley, – Sub-grantee PI MRC/UVRI/LSHTM Uganda Research Unit P.O. Box 49, Entebbe, Uganda Tel: ++256 774 778 869, Fax: +256 414 543002 E-mail: janet.seeley@lshtm.ac.uk janet.seeley@mrcuganda.org

Yunia Mayanja, Co-Investigator MRC/UVRI/ LSHTM Uganda Research Unit P.O. Box 49, Entebbe, Uganda E-mail: Yunia.Mayanja@mrcuganda.org

Elly Katabira Co-Investigator College of Health Sciences, Mulago Hospital Box 7072 Kampala, Uganda Tel: +256772401749

Victor Musiime, Co-Investigator College of Health Sciences, Mulago Hospital P.O. Complex, Box 7072 Kampala, Uganda Tel: +256772401749 E-mail: vmusiime@jcrc.org.ug

NIMH Grants Management Specialist:

NSC BG Rm 6138, 6001 Executive Blvd Rockville MD 20852, USA E-mail: rmunk@mail.nih.gov

# TABLE OF CONTENTS

| LIST OF ABBREVIATIONS | 4 |
|---|---|
| SUMMARY OF PROPOSED WORK | 5 |
| B. RATIONALE | 10 |
| C. AIMS | 11 |
| D. STUDY DESIGN AND METHODS | 12 |
| Overview of study design D.1 Study setting D.2 Intervention Components | |
| Intervention flow diagram | |
| D.3 Procedures - Phase 1 | 15 |
| D.3.1 Conduct facility site assessments | 15 |
| D.3.2 Qualitative data collection | |
| D.3.3 Operationalize curricula | |
| D.4 Phase 2; Pilot RCT | |
| D.4.1 Design of manuals and materials | |
| D.4.2 Standardize intervention materials | |
| D.4.3 Finalize study instruments and digital data collection forms | |
| D.4.4 Overview of Staff training | |
| D.4.5 Training Staff Counsellors/Mobilizers on HIV self-test | |
| D.4.6 Field test intervention | |
| D.4.7 Eligibility, screening and recruitment | |
| C.4.8 Randomization. | |
| D.4.9 Ethical Considerations | |
| D.4.10 Intervention Group Session Procedures | |
| D.4.11 PrEP Initiation and Monitoring. | |
| D.4.12 Follow-up Procedures. | |
| D.4.13 Training trial participants on HIV self-test | |
| D.4.14 Exit Interviews. | |
| D.4.15 Oral PrEP (Truvada) adherence counselling: | |
| D.5 Measures | |
| D.5.1 Primary outcome measurement | |
| D.5.2 Secondary Outcomes | |
| D.5.3 Mediators. | |
| D.6 Phase 3 | |
| D.7 Retention Plan | |
| D.8 Data quality and management | |
| D.9 Quantitative Data Analysis | |
| D.10 Qualitative Data Analysis | |
| E. SIGNIFICANCE OF THE PROPOSED WORK | |
| F. Timeline | 16 |

#### LIST OF ABBREVIATIONS

ANC Antenatal care

ART Antiretroviral therapy

ARV Antiretroviral

CAB Community Advisory Board

FGD Focus group discussion

FP Family planning
FSW Female sex worker
G/C Gonorrhea / chlamydia
GCP Good Clinical Practices

GHWP Good Health for Women Project

HIV ST HIV Self Test

HTC HIV testing and counseling IEC Independent Ethics Committee

IPV Interpersonal violence

IRB Institutional Review Board KII Key informant interview

LSHTM London School of Hygiene and Tropical Medicine

PCR Polymerase chain reaction

PE Peer educator

PMTCT Prevention of mother-to-child HIV transmission

PrEP Pre-exposure prophylaxis
RCT Randomized Controlled Trial
REC Research and Ethics Committee

SMS Short messaging system

SOC Standard of care

SOP Standard operating procedure SRH Sexual and reproductive health

sSA Sub-Saharan Africa

STI Sexually transmitted infection

UCSF University of California San Francisco

UNCST Uganda National Council for Science and Technology

UVRI Uganda Virus Research Institute

YAB Youth Advisory Board
YWHR Young women at high risk
WHO World Health Organization

## **SUMMARY OF PROPOSED WORK**

Background: Sub-Saharan Africa (sSA) is home to the fastest growing and youngest population in the world and includes countries with the highest HIV prevalence globally. More than half of sSA's population is under 25 years of age. Men and women aged 10-24, defined as 'young people' by the United Nations Population Fund (UNFPA), represent one third of the sSA population and this proportion continues to grow. Young sex workers, new to sex work, are much more vulnerable than their older colleagues to violence, STIs and HIV. The illegality of sex work in Uganda contributes to the risk these young women face. Effective STI and HIV prevention, care, support, and reproductive health services are critical to keeping this young vulnerable population healthy. Evidence on interventions that address uptake and adherence to HIV prevention services for high-risk populations is limited, and interventions that address young women at high risk (YWHR) are almost non-existent.

We propose to develop and conduct a pilot intervention trial including PrEP and HIV self-testing for HIV-uninfected women 15- to 24-years old who engage in high-risk sexual activity in Kampala, Uganda, and to evaluate its feasibility, acceptability and potential effect on PrEP uptake and adherence as well as repeat HIV self-testing. We will embed this study within our existing cohort study (NIMH R01 HD085805-01, PI King) that has revealed the need for greater attention to young sex workers soon after their initiation into the work. The intervention will focus on increasing initiation of PrEP among HIV-uninfected YWHR with enhanced adherence support, uptake of and adherence to repeat HIV self-test, and motivation to adopt and sustain sexual risk reduction behaviors for STI, HIV, and unplanned pregnancy.

Aims and Objectives: The main aim is to develop and assess an intervention to enhance initiation and adherence to PrEP among HIV negative YWHR. The specific aims are (1) To conduct formative research to enhance our understanding of the dynamics of the social and sexual networks, and context of young HIV-uninfected women (aged 15-24) engaged in high risk sexual behavior in Kampala, Uganda (2) Document barriers and opportunities for PrEP uptake and adherence as well as repeat HIV testing by self test; (3) To develop and test a socially and culturally acceptable and feasible prevention intervention on uptake and adherence to PrEP and HIV self-testing for young women at high risk for HIV; (4) to translate lessons learned from the pilot study to the design of a larger RCT.

#### A. BACKGROUND

Sub-Saharan Africa (sSA) is home to the fastest growing and youngest population in the world and includes countries with the highest HIV prevalence globally. More than half of sSA's population is under 25 years of age; men and women aged 10-24, defined as 'young people' by the United Nations Population Fund, represent one third of the sSA population and this proportion continues to grow.\(^1\)

Young women in sSA who are economically and educationally disadvantaged are at high risk of engaging in transactional sex. Transactional sex is a spectrum of economic interactions that varies from gift-giving to formal commercial sex work.<sup>2</sup> Factors such as age difference<sup>3</sup> and power disparity<sup>2,4,5</sup> between couples exist in most transactional sex situations. In some cases, sex work is the only source of family income, while in others, women use informal-transactional sex to supplement income or to augment social-status or material gain.<sup>6</sup> Transactional sex may be situational or temporary, associated with acute shortfalls in cash, need for school fees or food insecurity.<sup>2</sup> The prevalence of transactional sex varies by country and urban context in sSA,<sup>8</sup> with approximately 11.8% of girls and adolescent females reporting some exchange of sex for material goods in Uganda.<sup>9-11</sup>

Young women aged 15- to 24-years old involved in transactional sex work must be considered one of the highest risk populations in high HIV prevalence countries. 12.13 Globally, female sex workers (FSW) of all ages are over 10 times more likely to be infected with HIV than women in the general population. 14 In sSA in 2012, the average HIV prevalence among FSW was greater than 35%. 14 Throughout the world, 20-40% of sex workers enter sex work as adolescents with a mean age of entry of 16 years, and those under 16, new to sex work are much more vulnerable than their older colleagues to violence, STIs and HIV. 15-21 The illegality of sex work in Uganda further enhances the risk these young women face. Young people in Uganda have an HIV prevalence of 3.7% nationally, 22 yet young FSW have about a four to seven times higher prevalence of HIV. 22.23 Despite rising numbers of young FSW and their recognized vulnerability, there have been very few interventions globally that have targeted this group. 21

Adolescent and young women in Uganda are highly vulnerable to HIV, unplanned pregnancy and poor reproductive health outcomes. Adolescents are at especially high risk of maternal mortality, miscarriage and other complications in pregnancy.<sup>24</sup> Young Ugandans have less access to health services than adults, and even less so to HIV prevention

and care services.<sup>25</sup> Awareness of and knowledge about HIV transmission, reproductive health and contraceptive methods are poor among HIV-positive adolescents.<sup>10,11</sup> The large and growing population of young Ugandans face a range of social, economic, and health challenges,<sup>26,27</sup> yet their concerns may sometimes be overlooked in health agendas and programs.

This project is set within the Good Health for Women Project (GHWP), a study set up to investigate HIV and STI epidemiology and to enhance prevention strategies among women involved in high-risk sexual behavior in Kampala which has provided important data on the prevalence of HIV among this population and barriers faced by the young women engaged in high risk sexual activity. In 2011, the GHWP reported an HIV prevalence of 37%, among a cohort of 1,027 FSWs; of these, only 58% knew their HIV status at time of enrolment; 53% reported consistent condom use with paying clients in the last month.<sup>28</sup> Other studies have reported similar HIV prevalence and found young age to be a strong predictor of greater vulnerability to HIV, STI and violence. 15-21 28,29 GHWP results have shown high rates of STI, 30 the complexity and risks associated with sex work location, young age and FSW capacity to reduce harm, 6.29 how gender inequities have led to sex work and limited FSWs' ability to protect themselves. 31 Currently, GHWP participants 15-24 years old have an HIV prevalence of 28% and 24% report consistently using condoms. HIV incidence was 3.66/100 person-years (PY) and declined from 6.80/100PY in the first calendar year of the study enrollment. 29 HIV/AIDS is now the leading cause of death for women aged 15–29 years in sSA. 32-34 There is a dearth of evidence for effective interventions to increase HIV testing, prevention, adherence, retention in care amongst adolescents. 33,34 It is widely recognized that adolescents are difficult to reach as they often fall between pediatric and adult care. 35,36 To adequately reach youth, integrated structural, behavioral and biomedical, multi-level approaches will be required. Thus, combining biomedical approaches such as PrEP and HIV self-test with a prevention package, including behavioral and structural components as part of a comprehensive approach delivered by peers and counselors, could help to reduce HIV infection in young sex workers in diverse settings worldwide. 37

Trials among different high-risk populations have demonstrated high efficacy of tenofovir-based PrEP in reducing HIV transmission.  $\frac{38,39}{40}$  Thus, the 2015 WHO guidelines recommend PrEP for HIV-negative partners of HIV-infected individuals or populations engaged in high-risk behavior in settings with  $\geq 3\%$  annual HIV

incidence. 41. A recent study in South Africa and the US reported that adherence to daily PrEP is more difficult for younger populations, and low adherence was associated with decreased efficacy in all PrEP trials. 42 Barriers at the individual level included limited familiarity with antiretroviral-based prevention, stigma, storage, and social support, as well as structural hurdles including healthcare financing for PrEP, healthcare provider bias and ease with PrEP drugs, and the lack of youth-friendly health services. In its 2016 Consolidated Guidelines for HIV Prevention and Treatment, Uganda has approved PrEP for demonstration and pilot studies specifically for high-risk populations such as sex workers. 43

HIV self-testing (HIVST) was recommended by WHO in the 2014 comprehensive HIV care guidelines, and HIV testing guidelines from the Uganda Ministry of Health (2016), for use in demonstration projects. HIVST is defined as an individual performing and interpreting his/her own HIV test 44,45. It has the potential to be implemented at a wide scale with a minimal requirement for trained health-workers, and would thus be highly suited for FSW with low access to services. In addition, it is convenient since individuals perform HIVST in their own time, without having to present to a clinic at fixed hours. HIVST has been shown to be acceptable in a wide array of populations globally 46-54. It has recently been assessed in a number of settings in sub-Saharan countries, where it was found safe and accurate among the general population. Interest and acceptability in self-testing (HIV ST) is highest among high-risk groups 55-57. In Malawi, 92% of adult participants in a high prevalence setting opted for supervised self-testing over provider-delivered tests. 58 Respondents from a range of studies report that selftesting would reduce HIV testing stigma, a significant barrier to testing among young people. We will adapt a protocol that is being tested in Kenya among adult sex workers in Nairobi and Kisumu that found a high (98%) acceptance, gave accurate results and helped linkage to care. HIV ST could increase convenience and confidentiality, which are important testing barriers and can be especially useful for repeat testing in high HIV prevalence and incidence groups who may not visit health facilities regularly for long-term follow-up. 56,57,59,60 Repeat HIV self-tests can be empowering, can be a motivator to remain healthy and HIV-free, and can fit perfectly with PrEP. The Kenyan FSW study found that peers were able to assist with the tests, found no reports of harm, and that tests were empowering to users and can be cost-efficient. 61

Peer educators (PE) have an important role in health promotion for HIV prevention and PrEP. Numerous studies

have demonstrated that young people want information especially from trusted sources such as health care providers or teachers. 62.63 Acting as a bridge between communities and health facilities, Peer leaders and peer educators s can provide education, expedite access to the clinic, and promote adherence to health recommendations. Studies in Uganda have shown that community members view PE as knowledgeable and trustworthy in matters of health and would seek their advice if they had a medical problem. 64 Using peers in studies among young people have revealed that peer support as part of a comprehensive strategy to provide cognitive-behavioral counseling by a trusted adult has been effective. 65 Identifying effective strategies for improving uptake of adolescent HIV testing and re-testing for high risk groups 66 as well as successful uptake and adherence to effective prevention means including PrEP is critical for the survival of high risk youth and for the prevention of onward HIV transmission. This study could play a key role in understanding the complex connections between high risk sexual behavior, sexual relationship dynamics, socio-cultural relationship bargaining and sexual partnership decision-making that result in protected and unprotected sex in this highly vulnerable population. It will also help designing more effectively tailored interventions for HIV prevention and treatment for YWHR. Combining effective biomedical, behavioral and structural approaches is of key interest to Uganda's Ministry of Health as a potentially efficient way to reach marginalized populations at high risk for HIV acquisition. We propose to develop and pilot test a multicomponent intervention to improve uptake and adherence to PrEP and repeat HIV self-testing by HIV-negative YWHR 15- to 24-years old who are highly vulnerable to STI and HIV in Kampala, Uganda. We hypothesize that, combined with knowledge, skills and health-related self-efficacy, access to PrEP and HIV self-testing will act synergistically to prevent HIV and improve health outcomes of YWHR. Targeting young women who are initiating sex work will enable us to understand ways to enhance the potential impacts of a combined structural-behavioral intervention on health outcomes to be tested in a larger clinical trial. The study will provide important evidence to inform Uganda's HIV counseling and testing policy for adolescents and key populations, and will offer essential information for other countries striving for UNAIDS 90-90-90 target. In sum, this study could play a key role in understanding the complex connections between high-risk sexual behavior, sexual relationship dynamics, sociocultural relationship bargaining and sexual partnership decision-making that result in protected and unprotected sex in this highly vulnerable population. It will also help designing more effectively tailored interventions for HIV

prevention and treatment for YWHR.

#### **B. RATIONALE**

Targeting young Ugandan women at high risk for HIV (YWHR) and their social and sexual networks represents an innovation over traditional individual, partner or age-limited categories. Descriptive data that have been gathered on adolescent and young women engaged in high risk sexual activity in high HIV prevalence settings in sSA, though limited, reveal that they remain one of the most neglected, vulnerable, and underserved populations with regards to sexual and reproductive health (SRH) and HIV prevention services. 67,68

Combining the network and peer-led approaches that together put HIV combination prevention fully in control of women by using PrEP and repeat HIV self-tests may increase empowerment, acceptability, and penetration into networks and ultimately increase effectiveness in reaching this highly marginalized population. We believe it is key to focus our intervention on these women as soon as possible after they enter the sex trade in order to effect primary HIV prevention rather than wait until they attend the clinic after they may have already been infected. Preceding the design and pilot of our intervention with an in-depth qualitative formative phase will allow us to optimize the early identification of these women in their community, the delivery of interventions and the design of our study based on a more thorough understanding of the location, mobility and networks of young women at risk in Kampala.

We propose to use an innovative approach to linking HIV-negative YWHR to PrEP. Our participatory codesign approach is to engage YWHR in dialogue with researchers to co-develop intervention content and materials
that are responsive to the needs of the target group. We propose to use established co-design strategies to refine
aspects of the intervention and related materials to tailor them to our population. We will engage in conversation
young women who represent the intervention target population as well as individuals with biomedical, and program
expertise and experience with 'communities' who do not generally meet and discuss together. This participatory
design process will ensure YWHR the opportunity to engage meaningfully in designing an intervention that is
responsive to their needs and concerns.

Our study will be the first to use HIV self-tests for repeat testing among YWHR in sub-Saharan Africa. Few adolescent friendly services are available in Uganda, and stigma towards adolescent sexuality is pervasive among health workers. Self-test is a novel option that may allow a substantial proportion of these women to retest with the

help of a trained peer. There are limited data available on self-testing among similar groups, but what exists show a high level of acceptability<sup>69</sup> and low levels of social harm.<sup>70,71</sup>

HIV testing in urban hotspot areas will enhance effectiveness of these strategies in complex contexts and social environments, and will help overcome two key challenges of PrEP delivery; (1) identifying the most vulnerable communities to use PrEP and (2) enhancing adherence through repeat self-tests in a very high-risk population. It is premised on the hypothesis that offering acceptable strategies for HIV retesting by YWHR coupled with motivation to remain HIV negative through a peer-led community-engaged approach using a PrEP/repeat self test will empower YWHR to adopt risk reducing behavior.

## C. AIMS

We propose to design and refine key elements of our intervention components in order to maximize the probability of success in a definitive trial. The goal of the study is to develop and pilot test a multi-component structural and behavioral intervention targeting HIV-negative young women (15- to 24-years old) who engage in high-risk sexual activity in Kampala, Uganda, in order to increase uptake of, and adherence to combination HIV prevention services using PrEP, HIV self-tests, condoms and family planning. As currently conceptualized, the planned intervention will be delivered in two group sessions followed by two one-on-one counseling sessions. We will conduct the study in three integrated phases over 3 years:

Phase 1: will consist of formative research to enhance our understanding of barriers and opportunities for PrEP and HIV testing uptake and adherence as well as to better understand the dynamics of the social and sexual networks, mobility and context of young women (15- to 24-years old) engaged in high risk sexual behavior in Kampala, Uganda. In our current R01 study (A Cognitive Behavioral And Structural HIV Prevention Intervention for Young Ugandan Sex Workers) we have found that hot spots are not static and must be identified regularly with the input of key informants who are peers of our target population. We will collect qualitative data using in-depth interviews and focus group discussions with key stakeholders: a) HIV-positive YWHR, b) HIV-negative YWHR, c) male partners of YWHR, d) peer educators, e) health workers and f) policy makers (including ministry of health officials). The objective of these discussions will be to identify the opportunities and multiple levels of barriers to specific HIV prevention services as well as the acceptability, feasibility, challenges to our preliminary intervention

components (Table 1). We will examine our planned approach with respect to social and cultural relevance as well as necessary resources, and how to operationalize the intervention components most efficiently considering existing services, the knowledge, capacity and attitudes of potential participants, as well as the different contexts they are living in (eg cramped shared housing; high mobility). We will use participatory co-design methods to produce and pilot a training curriculum and associated materials for use in intervention group sessions. These materials will be refined with input from a youth advisory board (YAB) in a second series of focus group discussions with members of the target population.

<u>Phase 2:</u> Will be informed by Phase 1. We will conduct a small pilot RCT study (N=60) to assess the feasibility, acceptability, and preliminary effects of the intervention on PrEP uptake and adherence.

<u>Phase 3</u>: We will review qualitative and quantitative data on intervention feasibility, acceptability and potential effectiveness from Phase 2 in collaboration with the Community Advisory Board (CAB) and Youth Advisory Board (YAB) to seek consensus about refinements to be made for formulating an R01 application to assess the efficacy of the intervention in a larger RCT. The setting, conceptual framework and activities of each phase are described below.

# D. STUDY DESIGN AND METHODS

#### **OVERVIEW OF STUDY DESIGN**

In this pilot study, we propose to conduct formative research and then develop and evaluate a combination prevention intervention through a randomized controlled trial comparing intervention vs GHWP care among high-risk young people.



## **D.1 Study setting**

We will conduct this study at the GHWP Clinic in Kampala. The GHWP clinic is located in a densely populated slum area of southern Kampala with retail shops and roadside kiosks selling general merchandise, and bars, which are the main hotspots in the area. The current HIV prevalence among women in the cohort who are 15-24 years is about 31% and 38% in all participants. The GHWP clinic currently provides mobilization, testing and counseling, and ART. 28.72 At GHWP, all eligible participants receive HIV care and treatment, including ART, in accordance with Uganda MoH Guidelines. Peer educators associated with the clinic visit YWHR to provide information, education and referral related to uptake and retention to clinic services according to established visit protocols. The existing GHWP infrastructure, highly skilled staff, and proven recruitment system 31.73.74 are strong assets to this study. Participants will be recruited from hotspots (generally bars and lodges) in Kampala according to established and tested protocols. The clinic currently provides free medical and counseling services, free male and female condoms, HIV and STI testing and treatment to all high risk women, their partners and their children under 5 years

of age. GHWP has over 4358 enrolled FSW, 36% of whom are under 24 years of age, and enrolment is open and ongoing. However, currently there are limited specialized services for *young* women engaged in some form of transactional sex at GHWP apart from our parent study (NIMH R01 HD085805-01 PI King) and neither PrEP nor HIV self-testing are currently offered as standard services.

# **D.2 Intervention Components**

The content and structure of the intervention will include at a minimum 2 group sessions and 2 counseling sessions with YWHR (Table 1), which will be facilitated by trained peers and counselors. Group sessions will be limited to 8 participants, last about 2- 3 hours, be participatory, youth-centered and include modeling, role plays, story-telling, and body-mapping – all strategies that we have previously found to be highly engaging with young people and lower literacy populations. As our population has low literacy, our techniques will be highly visual to ensure accessibility to information and avoid stigmatizing participants who cannot read. Sessions will be conducted in Luganda and/or English at the clinic, as it is comfortable and private and is where we conduct the intervention for our current R01. The clinicians will be blinded to the intervention. Google mapping of hotspots will be done at every scheduled visit. This intervention format will be revised based on findings of Phase 1 formative research

#### INTERVENTION FLOW DIAGRAM

# **Table 1: Intervention Components**

**Screening:** HIV counseling and testing either in the community hot spots or in the clinic followed by: **TWO GROUP SESSIONS** covering multi-level factors *informed by formative phase and parent study*:

- 1. <u>Health empowerment</u>: Barriers and strategies for health seeking, benefits, process and efficacy of PrEP, adherence support guidance, safer sex, HIV and reproductive health including STI prevention and treatment, family planning, child spacing & contraceptive methods; *Curriculum to be drawn from existing resources (current R01 + PrEP demonstration project; Dr Katabira)*
- 2. <u>Initiating daily PrEP</u> following MOH guidelines (300mg TDF + 200mg FTC)
- 3. <u>Social/Contextual empowerment</u>: building a support network using SMS reminders designed by peers from parent study; focusing on gender and social norms; training in HIV self-testing; exploring issues around education and life ambitions, vocational training and alternative livelihoods; *To be drawn/adapted from existing curricula*

## TWO INDIVIDUAL COUNSELING SESSIONS covering:

Personal history; cognitive behavioral therapy (CBT) as relevant; HIV/STI transmission risk at multiple levels; Uptake of PrEP, safer sex, family planning, violence prevention; Adherence to PrEP, safer sex, family planning, clinic visits; Remaining HIV negative: re-testing using HIV self-test; Exploring education and life ambitions, and alternative livelihoods

#### **D.3 Procedures - Phase 1**

D.3.1 Conduct facility site assessments to assist future randomization procedures and power calculations.

As part of Phase 1 and during the first year of the R34 project, a field team will conduct detailed mapping of all current hot spots for young women in urban Kampala including areas where high-risk youth congregate with their social networks. Ten communities with separate catchment areas and similar baseline characteristics will be identified as study sites (for the future R01 application) through qualitative and quantitative data collection using a mapping protocol that we have used in previous studies. 25 Briefly, this protocol involves showing the participant a map of Kampala on Google-Maps and them pinning their hotspot(s). In-depth and key informant interviews and focus group discussions will assess acceptability, feasibility, challenges and potential uptake of the proposed strategies. We will examine the social and cultural relevance and how to operationalize the procedures considering the knowledge, attitudes and context of the target population. The maps will be kept highly confidential and anonymous in a locked cabinet in the study office. Only study IDs will be used; no names and no telephone numbers will be connected to study participant information. In addition, we will collect information on predefined criteria (e.g. number and ages of potential participants at a given hotspot at the time of the visit, willingness to be enrolled, location, description of site [e.g., bar, lodge], and availability of space suitable for outreach testing). Site assessments will also serve as an opportunity for mobilization team to familiarize themselves fully for a smooth transition from the pilot to the proposed RCT. A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This web site will not include information that can identify the participant. At most, the web site will include a summary of the results.

D.3.2 Qualitative data collection on risk, barriers to HIV prevention services and intervention content.

**Table 2: Qualitative Data Collection** 

| Group | | Topic | Method | # participants |
|---|---|---|---|---|
| | Risk | Intervention | | |
| HIV negative YWHR | Х | Х | FGD, | 8x2= 16 |
| | | | Interviews | 8 |
| HIV positive YWHR | Х | Х | FGD, | 1x8=8 |
| · | | | Interviews | 8 |
| Peer educators | | Х | FGD | 8 |
| Male partners | Х | | FGD | 8 |
| Key Informants (health | | Х | Interviews | 8 |
| workers, policy makers) | | | | |
| TOTAL | | | | 64 |

Focus group discussions will be organized with HIV negative and positive YWHR, Peer Educators, male partners and other key stakeholders (Table 2) to inform the content and form of the intervention group discussions. The discussions will be held in the clinic and notes will be taken immediately. With YWHR, discussions will assess both the areas of risk behavior and barriers to accessing HIV prevention services as well as feasibility, acceptability and refinement of the intervention design and materials to be used in the next phase as well as documenting most relevant strategies for the target group. Discussions will focus on possible pathways of effectiveness such as

knowledge, social support, motivation and skills. With PE and other key informants, the discussion will focus on topics surrounding how to develop and implement the intervention in the most effective, targeted manner. With YWHR, PE and key informants, we will explore the following alternatives to simple self-report through group discussions and interviews with participants:

- 1) Assisted ST; at the time of receiving the HIV ST, participants will be offered to perform it in the presence of their counselor who can then directly counsel the participant according to her questions and/or test result
- 2) Delivery of the HIV self-test (ST) result strip into a labeled box just inside the clinic gate; each HIV ST strip will have a bar code on it and participants can drop their strip into the box as they enter or exit the clinic. At enrolment, these procedures would be explained in detail
- 3) Participants with phones can report their HIV ST experience on a four-question phone-based short messaging system (SMS) survey: (Did you use your test? Was it easy or difficult? Would you use it again? Would you like help?) and upload their responses into a simple web-based portal. We are using web-based portals in other studies as well as on a national level for Ugandan PMTCT data entry and the development and use of the portal have proven simple, user-friendly and functional <sup>76</sup>.

# D.4 Phase 2; Pilot RCT

The pilot RCT will assess intervention feasibility/acceptability and control conditions to be used in a subsequent larger trial. We will examine preliminary impact on mediators and outcomes of interest.

#### F. TIMELINE

Table 6: Outline of Project Activities by Year and Quarter

| | Year 1<br>Oct 17-Sept 18 | | | Year 2<br>Oct 18-Sept 19 | | | Year 3<br>Oct 19-Sept 20 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activities Quarter | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 |
| Planning & staff recruitment; Assemble YAB, | | | | | | | | | | | | |
| Phase 1: Formative research | | | | | | | | | | | | |
| Phase 2: Screening & enrolment Pilot Study | | | | | | | | | | | | |
| Phase 2: Follow-up Pilot | | | | | | | | | | | | |
| Phase 2: Analysis | | | | | | | | | | | | |
| Phase 3: Translate results (feasibility and | | · | · | | | · | · | | | | | |

#### REFERENCES

- 1. UNFPA. Adolescents and Young People in Sub-Saharan Africa Opportunities and Challenges. Johannesburg: UNFPA;2012.
- 2. MacPherson EE, Sadalaki J, Njoloma M, et al. Transactional sex and HIV: understanding the gendered structural drivers of HIV in fishing communities in Southern Malawi. *J Int AIDS Soc.* Jun 14 2012;15 Suppl 1:1-9.
- 3. Ngugi EN, Benoit C, Hallgrimsdottir H, Jansson M, Roth EA. Family Kinship Patterns and Female Sex Work in the Informal Urban Settlement of Kibera, Nairobi, Kenya. *Hum Ecol Interdiscip J.* Jun 2012;40(3):397-403.
- 4. Dunkle KL, Jewkes RK, Brown HC, Gray GE, McIntryre JA, Harlow SD. Gender-based violence, relationship power, and risk of HIV infection in women attending antenatal clinics in South Africa. *Lancet*. May 01 2004;363(9419):1415-1421.
- 5. Jewkes RK, Dunkle K, Nduna M, Shai N. Intimate partner violence, relationship power inequity, and incidence of HIV infection in young women in South Africa: a cohort study. *Lancet*. Jul 03 2010;376(9734):41-48.
- 6. Mbonye M, Nakamanya S, Nalukenge W, King R, Vandepitte J, Seeley J. 'It is like a tomato stall where someone can pick what he likes': structure and practices of female sex work in Kampala, Uganda. *BMC Public Health*. Aug 10 2013;13:741.
- 7. Miller CL, Bangsberg DR, Tuller DM, et al. Food insecurity and sexual risk in an HIV endemic community in Uganda. *AIDS Behav*. Oct 2011;15(7):1512-1519.
- 8. Konde-Lule JK, Sewankambo N, Morris M. Adolescent sexual networking and HIV transmission in rural Uganda. *Health Transit Rev.* 1997;7 Suppl:89-100.
- 9. Walker D, Pereznieto, P, Bantebya, G, Ochen, E. Sexual exploitation of adolescent girls in Uganda: The drivers, consequences and responses to the 'sugar daddy' phenomenon. Kampala, Uganda: ODI;2014.
- 10. Bakeera-Kitaka S, Nabukeera-Barungi N, Nostlinger C, Addy K, Colebunders R. Sexual risk reduction needs of adolescents living with HIV in a clinical care setting. *AIDS Care*. Apr 2008;20(4):426-433.
- 11. Lowenthal ED, Bakeera-Kitaka S, Marukutira T, Chapman J, Goldrath K, Ferrand RA. Perinatally acquired HIV infection in adolescents from sub-Saharan Africa: a review of emerging challenges. *Lancet Infect Dis.* Jul 2014;14(7):627-639.
- 12. Idele P, Gillespie A, Porth T, et al. Epidemiology of HIV and AIDS among adolescents: current status, inequities, and data gaps. *J Acquir Immune Defic Syndr*. Jul 01 2014;66 Suppl 2:S144-153.
- 13. Stover J, Rosen J, Kasedde S, Idele P, McClure C. The impact and cost of the HIV/AIDS investment framework for adolescents. *J Acquir Immune Defic Syndr*. Jul 01 2014;66 Suppl 2:S170-175.
- 14. Baral S, Beyrer C, Muessig K, et al. Burden of HIV among female sex workers in low-income and middle-income countries: a systematic review and meta-analysis. *Lancet Infect Dis.* Jul 2012;12(7):538-549.
- 15. Goldenberg S, Silverman J, Engstrom D, Bojorquez-Chapela I, Strathdee S. "Right Here is the Gateway": Mobility, Sex Work Entry and HIV Risk Along the Mexico-U.S. Border. *Int Migr.* Aug 01 2014;52(4):26-40.
- 16. Goldenberg SM, Chettiar J, Simo A, et al. Early sex work initiation independently elevates odds of HIV infection and police arrest among adult sex workers in a Canadian setting. *J Acquir Immune Defic Syndr*. Jan 01 2014;65(1):122-128.
- 17. Goldenberg SM, Rangel G, Vera A, et al. Exploring the impact of underage sex work among female sex workers in two Mexico-US border cities. *AIDS Behav.* May 2012;16(4):969-981.
- 18. Odinokova V, Rusakova M, Urada LA, Silverman JG, Raj A. Police sexual coercion and its association with risky sex work and substance use behaviors among female sex workers in St. Petersburg and Orenburg, Russia. *Int J Drug Policy*. Jan 2014;25(1):96-104.

- 19. Rocha-Jimenez T, Brouwer KC, Silverman JG, Morales-Miranda S, Goldenberg SM. Exploring the Context and Implementation of Public Health Regulations Governing Sex Work: A Qualitative Study with Migrant Sex Workers in Guatemala. *J Immigr Minor Health*. Mar 25 2016.
- 20. Servin AE, Brouwer KC, Gordon L, et al. Vulnerability Factors and Pathways Leading to Underage Entry into Sex Work in two Mexican-US Border Cities. *J Appl Res Child*. 2015;6(1).
- 21. Silverman JG. Adolescent female sex workers: invisibility, violence and HIV. *Arch Dis Child.* May 2011;96(5):478-481.
- 22. MOH. Uganda AIDS Indicator Survey 2011. Kampala, Uganda and Calverton, Maryland, USA2012.
- 23. MOH. *The Crane Survey Report*. Kampala, Uganda: MOH;2009.
- 24. Bearinger LH, Sieving RE, Ferguson J, Sharma V. Global perspectives on the sexual and reproductive health of adolescents: patterns, prevention, and potential. *Lancet*. Apr 07 2007;369(9568):1220-1231.
- 25. WHO. Global Update on HIV Treatment 2013: Results, Impact and Opportunities. Geneva: WHO;2013.
- 26. UNICEF. Children in an Urban World. New York, NY: UNICEF;2012.
- 27. UNICEF. The State of the World's Children 2014: Every Child Counts. 2014; <a href="http://www.unicef.org/sowc2014/numbers/documents/english/EN-FINAL FULL REPORT.pdf">http://www.unicef.org/sowc2014/numbers/documents/english/EN-FINAL FULL REPORT.pdf</a>.
- 28. Vandepitte J, Bukenya J, Weiss HA, et al. HIV and other sexually transmitted infections in a cohort of women involved in high-risk sexual behavior in Kampala, Uganda. *Sex Transm Dis.* 2011;38(4):316-323.
- 29. Vandepitte J, Weiss HA, Bukenya J, et al. Alcohol use, mycoplasma genitalium, and other STIs associated With HIV incidence among women at high risk in Kampala, Uganda. *J Acquir Immune Defic Syndr*. Jan 1 2013;62(1):119-126.
- 30. Vandepitte J, Muller E, Bukenya J, et al. Prevalence and correlates of Mycoplasma genitalium infection among female sex workers in Kampala, Uganda. *J Infect Dis.* Jan 15 2012;205(2):289-296.
- 31. Mbonye M, Nalukenge W, Nakamanya S, et al. Gender inequity in the lives of women involved in sex work in Kampala, Uganda. *J Int AIDS Soc.* Jun 14 2012;15 Suppl 1:1-9.
- 32. Crankshaw TL, Voce A, King RL, Giddy J, Sheon NM, Butler LM. Double disclosure bind: complexities of communicating an HIV diagnosis in the context of unintended pregnancy in Durban, South Africa. *AIDS Behav.* Jan 2014;18 Suppl 1:S53-59.
- 33. Buzdugan R, Copas A, Moses S, et al. Devising a female sex work typology using data from Karnataka, India. *Int J Epidemiol*. Apr 2010;39(2):439-448.
- 34. Buzdugan R, Halli SS, Cowan FM. The female sex work typology in India in the context of HIV/AIDS. *Trop Med Int Health.* Jun 2009;14(6):673-687.
- 35. Cluver LD, Orkin FM, Yakubovich AR, Sherr L. Combination Social Protection for Reducing HIV-Risk Behavior Among Adolescents in South Africa. *J Acquir Immune Defic Syndr*. May 01 2016;72(1):96-104.
- 36. Toska E, Gittings L, Hodes R, et al. Resourcing resilience: social protection for HIV prevention amongst children and adolescents in Eastern and Southern Africa. *Afr J AIDS Res.* Jul 2016;15(2):123-140.
- 37. Bekker LG, Johnson L, Cowan F, et al. Combination HIV prevention for female sex workers: what is the evidence? *Lancet*. Jan 03 2015;385(9962):72-87.
- 38. Baeten JM, Donnell D, Ndase P, et al. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. *N Engl J Med.* Aug 2 2012;367(5):399-410.
- 39. Grant RM, Lama JR, Anderson PL, et al. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. *N Engl J Med.* Dec 30 2010;363(27):2587-2599.
- 40. Carrion A, Miles, J, Mosley, J, . Prevention Strategies Against HIV Transmission
- A Proactive Approach. Journal of Pharmacy Practice. 2017.
- 41. WHO. Guideline on when to start antiretroviral therapy and on pre-exposure prophylaxis for HIV. Geneva: WHO;2015.
- 42. Hosek S, Celum C, Wilson CM, Kapogiannis B, Delany-Moretlwe S, Bekker LG. Preventing HIV among adolescents with oral PrEP: observations and challenges in the United States and South Africa. *J Int AIDS Soc.* 2016;19(7(Suppl 6)):21107.
- 43. MOH. Consolidated Guidelines for Prevention and Treatment of HIV in Uganda2016.
- 44. Lippman SA, Moran L, Sevelius J, et al. Acceptability and Feasibility of HIV Self-Testing Among Transgender Women in San Francisco: A Mixed Methods Pilot Study. *AIDS Behav*. Apr 2016;20(4):928-938.

- 45. Volk JE, Lippman SA, Grinsztejn B, et al. Acceptability and feasibility of HIV self-testing among men who have sex with men in Peru and Brazil. *Int J STD AIDS*. Jun 2016;27(7):531-536.
- 46. Tucker JD, Wei C, Pendse R, Lo YR. HIV self-testing among key populations: an implementation science approach to evaluating self-testing. *Journal of virus eradication*. Jan 2015;1(1):38-42.
- 47. Volk JE, Lippman SA, Grinsztejn B, et al. Acceptability and feasibility of HIV self-testing among men who have sex with men in Peru and Brazil. *International journal of STD & AIDS*. May 12 2015.
- 48. Figueroa C, Johnson C, Verster A, Baggaley R. Attitudes and Acceptability on HIV Self-testing Among Key Populations: A Literature Review. *AIDS and behavior*. Jun 9 2015.
- 49. Wood BR, Ballenger C, Stekler JD. Arguments for and against HIV self-testing. *Hiv/Aids*. 2014;6:117-126.
- 50. Young SD, Daniels J, Chiu CJ, et al. Acceptability of using electronic vending machines to deliver oral rapid HIV self-testing kits: a qualitative study. *PloS one*. 2014;9(7):e103790.
- 51. Wong V, Johnson C, Cowan E, et al. HIV self-testing in resource-limited settings: regulatory and policy considerations. *AIDS and behavior*. Jul 2014;18 Suppl 4:S415-421.
- 52. Kalibala S, Tun W, Cherutich P, Nganga A, Oweya E, Oluoch P. Factors associated with acceptability of HIV self-testing among health care workers in Kenya. *AIDS and behavior*. Jul 2014;18 Suppl 4:S405-414.
- 53. Krause J, Subklew-Sehume F, Kenyon C, Colebunders R. Acceptability of HIV self-testing: a systematic literature review. *BMC public health*. 2013;13:735.
- 54. Ng OT, Chow AL, Lee VJ, et al. Accuracy and user-acceptability of HIV self-testing using an oral fluid-based HIV rapid test. *PloS one*. 2012;7(9):e45168.
- 55. NASCOP. National AIDS and STD Control Programme, Preparedness for HIV/AIDS service delivery: The 2005 Kenya Health Workers Survey. In: Ministry of Health Kenya, ed. Nairobi: NASCOP; 2006.
- 56. Carballo-Dieguez A, Frasca T, Dolezal C, Balan I. Will gay and bisexually active men at high risk of infection use over-the-counter rapid HIV tests to screen sexual partners? *Journal of sex research*. 2012;49(4):379-387.
- 57. Lee VJ, Tan SC, Earnest A, Seong PS, Tan HH, Leo YS. User acceptability and feasibility of self-testing with HIV rapid tests. *Journal of acquired immune deficiency syndromes* (1999). Aug 1 2007;45(4):449-453.
- 58. Choko A, Desmond N, Webb E, et al. The Uptake and Accuracy of Oral Kits for HIV Self-Testing in High HIV Prevalence Setting: A Cross-Sectional Feasibility Study in Blantyre, Malawi. *PLoS medicine*, 2011. 2011;8(10):p. e1001102.
- 59. Gaydos CA, Hsieh YH, Harvey L, et al. Will patients "opt in" to perform their own rapid HIV test in the emergency department? *Annals of emergency medicine*. Jul 2011;58(1 Suppl 1):S74-78.
- 60. Sharma A, Sullivan PS, Khosropour CM. Willingness to Take a Free Home HIV Test and Associated Factors among Internet-Using Men Who Have Sex with Men. *Journal of the International Association of Physicians in AIDS Care (Chicago, Ill. : 2002)*. Nov-Dec 2011;10(6):357-364.
- 61. Mavedzenge N, Baggaley R, Corbett EL. A review of self-testing for HIV: research and policy priorities in a new era of HIV prevention. *Clin Infect Dis.* Jul 2013;57(1):126-138.
- 62. Guttmacher. Protecting the Next Generation in Sub-Saharan Africa: Learning from Adolescents to Prevent HIV and Unintended Pregnancy. 2007.
- 63. WHO. Adolescent Friendly Health Services An Agenda for Change. Geneva: WHO;2002.
- 64. Mitchell K, Nakamanya S, Kamali A, Whitworth JA. Community-based HIV/AIDS education in rural Uganda: which channel is most effective? *Health Educ Res.* Aug 2001;16(4):411-423.
- 65. Swahn MH, Braunstein S, Kasirye R. Demographic and psychosocial characteristics of mobile phone ownership and usage among youth living in the slums of Kampala, Uganda. *West J Emerg Med.* Aug 2014;15(5):600-603.
- 66. MOH. *National Implementation Guidelines for HIV Counselling and Testing in Uganda*. Kampala, Uganda: Uganda Ministry of Health;2010.
- 67. World Health Organization. *HIV and adolescents: guidance for HIV testing and counselling and care for adolescents living with HIV.* Geneva: World Health Organization; 2013.
- 68. UNAIDS. The GAP Report 2014: UNAIDS, Geneva, Switzerland; 2014.
- 69. Pant Pai N, Sharma J, Shivkumar S, et al. Supervised and unsupervised self-testing for HIV in high- and low-risk populations: a systematic review. *PLoS Med.* 2013;10(4):e1001414.

- 70. Thirumurthy H, Masters SH, Mavedzenge SN, Maman S, Omanga E, Agot K. Promoting male partner HIV testing and safer sexual decision making through secondary distribution of self-tests by HIV-negative female sex workers and women receiving antenatal and post-partum care in Kenya: a cohort study. *Lancet HIV*. Jun 2016;3(6):e266-274.
- 71. Choko AT, Desmond N, Webb EL, et al. The uptake and accuracy of oral kits for HIV self-testing in high HIV prevalence setting: a cross-sectional feasibility study in Blantyre, Malawi. *PLoS Med.* Oct 2011;8(10):e1001102.
- 72. Mbonye M, Seeley J, Nalugya R, et al. Test and treat: the early experiences in a clinic serving women at high risk of HIV infection in Kampala. *AIDS Care*. 2016;28 Suppl 3:33-38.
- 73. Seeley J, Russell S, Khana K, Ezati E, King R, Bunnell R. Sex after ART: sexual partnerships established by HIV-infected persons taking anti-retroviral therapy in Eastern Uganda. *Culture, health & sexuality*. Oct 2009;11(7):703-716.
- 74. Vandepitte J WH, Bukenya J, Nakubulwa S, Mayanja Y, Matovu G, Kyakuwa N,Hughs P, Hayes R, Grosskurth, H. Alcohol use, Mycoplasma genitalium and other STIs associated with HIV incidence among women at high risk in Kampala, Uganda. *JAIDS*. 2013;62(1)(1):119-126.
- 75. Hladik W, Sande, E, Bogere, T, Borders, S, Opio, A, Tobiasa, J. Survey-informed mapping and localized size estimation of key populations at increased risk of HIV infection in Kampala, Uganda. *Draft Manuscript*. 2016.
- 76. Radin AK, Abutu AA, Okwero MA, et al. Confronting Challenges in Monitoring and Evaluation: Innovation in the Context of the Global Plan Towards the Elimination of New HIV Infections Among Children by 2015 and Keeping Their Mothers Alive. *J Acquir Immune Defic Syndr*. May 01 2017;75 Suppl 1:S66-S75.
- 77. Earle KE, Seneviratne T, Shaker J, Shoback D. Fanconi's syndrome in HIV+ adults: report of three cases and literature review. *J Bone Miner Res.* May 2004;19(5):714-721.
- 78. Wilson I LY, Michaud J, Fowler F, Jr and Rogers W. Validation of a new three-item self-report measure for medication adherence. *AIDS Behav.* 2016.
- 79. MOH. Adolescent Health Policy Guidelines and Service Standards for Uganda. Uganda: MOH2011.
- 80. MOH. Adolescent Sexual and Reproductive Health: A Job Aide 2012. 2012.
- 81. Evans D MC, Mahomed K, et al. Treatment outcomes of HIV-infected adolescents attending public-sector HIV clinics across Gauteng and Mpumalanga, South Africa. *AIDS research and human retroviruses*. 2013;29:892-900.
- 82. Gelberg L AR, Leake BD. The Behavioral Model for Vulnerable Populations: application to medical care use and outcomes for homeless people. *Health services research*. 2000;34:1273-1302.
- 83. Pulerwitz J GS, DeJong W,. Measuring sexual relationship power in HIV/STD research. *Sex Roles*. 2000;42(7):637-660.
- 84. Straus M HS, Boney-McCoy S, Sugarman D. Measuring sexual relationship power in HIV/STD research. *J Fam Issues*. 1996;17(3):283-316.
- 85. Derogatis LR, Lipman RS, Rickels K, Uhlenhuth EH, Covi L. The Hopkins Symptom Checklist (HSCL). A measure of primary symptom dimensions. *Mod Probl Pharmacopsychiatry*. 1974;7(0):79-110.
- 86. Bolton P, Wilk CM, Ndogoni L. Assessment of depression prevalence in rural Uganda using symptom and function criteria. *Soc Psychiatry Psychiatr Epidemiol*. Jun 2004;39(6):442-447.
- 87. Erlen JA CE, Kim KH, Caruthers D and Sereika SM. The HIV Medication Taking Self-efficacy Scale: Psychometric evaluation. *J Adv Nurs*. 2010;66(11):2560-2572.
- 88. Pronyk PM, Hargreaves JR, Kim JC, et al. Effect of a structural intervention for the prevention of intimate-partner violence and HIV in rural South Africa: a cluster randomised trial. *Lancet*. Dec 2 2006;368(9551):1973-1983.
- 89. Hu Y, Lu H, Raymond HF, et al. Measures of condom and safer sex social norms and stigma towards HIV/AIDS among Beijing MSM. *AIDS Behav*. Jun 2014;18(6):1068-1074.
- 90. Bradley KA DA, Volk RJ, Williams EC, Frank D, Kivlahan DR. AUDIT-C as a brief screen for alcohol misuse in primary care. *Alcoholism, clinical and experimental research*. 2007;31:1208-1217.
- 91. Apondi R BR, Awor A, . Home-based antiretroviral care is associated with positive social outcomes in a prospective cohort in Uganda. *Journal of acquired immune deficiency syndromes*. 2007;44:71-76.

- 92. Broadhead WE GS, de Gruy FV, Kaplan BH. T. The Duke-UNC Functional Social Support Questionnaire. Measurement of social support in family medicine patients. *Medical care*. 1988;26:709-723.
- 93. Little R, Rubin D. Statistical Analysis with Missing Data. New York: John Wiley & Sons; 1987.
- 94. Gertler P.J., Martinez S, Premand P, Rawlings LB, Vermeersch CMJ. *Impact Evaluation in Practice*. Washington DC: he International Bank for Reconstruction and Development / The World Bank;;2011.
- 95. Richie J, Spencer L, eds. Analyzing Qualitative Data. London: Routeledge; 1994.
- 96. Thorne S. *Interpretive Description*. Vol 2. Walnut Creek, Ca: Left Coast Press, Inc.; 2008.
- 97. Creswell J. *Qualitative Inquiry & Research Design: Choosing Among Five Approaches*. Second Edition ed. Thousand Oaks: Sage Publications; 2007.